CLINICAL TRIAL: NCT01681511
Title: A Randomized Trial for the Safety and Effectiveness of a Novel Antimicrobial-Coated Foley Catheter Attached to an Antimicrobial Anti-Reflux Device for Reduction of Catheter-Associated Urinary Tract Infection
Brief Title: A Trial for the Safety and Effectiveness of a Novel Antimicrobial-Coated Foley Catheter for Reduction of CAUTI.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Innovative Chemical and Environmental Technologies, Inc (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ICET-001; R44DK055891-06 (NIH)
Record Dates: First submitted 2012-07-29; First posted 2012-09-10 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Urinary Tract Infection
Keywords: Catheter Associated Urinary Tract Infections; CAUTI
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICET™ TIC Foley Catheter (Experimental): Route of Administration: Urinary Bladder Catheterization
  Interventions: Device: ICET™ TIC Foley Catheter
- BARD® LUBRI-SIL® IC Foley Catheter (Active Comparator): Route of Administration: Urinary Bladder Catheterization
  Interventions: Device: BARD® LUBRI-SIL® IC Foley Catheter

INTERVENTIONS:
Device: ICET™ TIC Foley Catheter — The device to be evaluated in this investigation is a silver-based antimicrobial coated Foley catheter connected to an antimicrobial anti-reflux accessory (ICET Inc, Norwood, MA). The closed system is referred to as the TIC system and is designed with the objective of reducing the incidence of CAUTI. The accessory is non-tissue contacting.
  Other Names: ICET™ TIC Foley Catheter Device (TIC System)
  Arms: ICET™ TIC Foley Catheter
Device: BARD® LUBRI-SIL® IC Foley Catheter — The LUBRI-SIL® I.C. antimicrobial 100% silicone Foley catheter incorporates a formulation consisting of BACTI-GUARD®* silver alloy coating and BARD® hydrogel.
  Other Names: BARD ® LUBRI-SIL® I.C. Foley Catheter Device
  Arms: BARD® LUBRI-SIL® IC Foley Catheter

SUMMARY:
The primary objective of this pilot study is to demonstrate the feasibility of recruiting eligible patients for the purposes of assessing the temporal aspects and rates of Catheter Associated Urinary Tract Infection (CAUTI), based on the agreed-upon case definition so that the numbers needed for a pivotal study can be better estimated.

DETAILED DESCRIPTION:
This pilot study will be a prospective, single site, randomized clinical investigation comparing the safety and effectiveness of the ICET TIC antimicrobial Foley catheter, against the infection control standard-of-care, the BARD ® LUBRI-SIL® I.C. Foley catheter.

Approximately 160 patients will be screened. The study has been designed to enroll approximately 120 eligible subjects to obtain about 60 evaluable subjects (30 in each arm). Subjects who meet the eligibility criteria will be enrolled into the study and randomly assigned to the experimental or standard-of-care group in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Subject is expected to be catheterized with 14 or 16 French Foley catheters for at least 72 hours.
3. Subject (or a legally authorized representative) has provided written informed consent for study participation and procedures to be performed.
4. Life expectancy at least 3 months or more in the judgment of the investigator

Exclusion Criteria:

1. Subjects who present with previously known, symptomatic UTI
2. Subjects with a positive urine dipstick at the time of enrollment
3. Subjects who are on systemic antibiotics within 48 hours prior to enrollment
4. Subjects with a known of suspected allergy to silicone, silver or silver compounds causing delayed hypersensitivity reactions or contact dermatitis.
5. Subjects who have had an indwelling catheter removed less than 48 hours before study enrollment.
6. Current genitourinary tract surgery or known infection
7. Subject requires use of a non-study urinary catheter
8. Subjects known to be pregnant or breast feeding at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Kline, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Fairview medical center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Leuck AM, Johnson JR, Hunt MA, Dhody K, Kazempour K, Ferrieri P, Kline S. Safety and efficacy of a novel silver-impregnated urinary catheter system for preventing catheter-associated bacteriuria: a pilot randomized clinical trial. Am J Infect Control. 2015 Mar 1;43(3):260-5. doi: 10.1016/j.ajic.2014.11.021. PMID 25728152

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single Site Recruitment
Pre-assignment Details: As of Study Termination: 100 Sbj signed Informed Consent, 95 Sbj RND
  Definitions:
  Safety Pop=Any Sbj receiving treatment after RND
  Evaluable Pop=All RND Sbj successfully CZD ≥ 72±24 hours w/out systemic (post-op) antibiotic for CZD/non-CZD related reasons.
  CZD=catheterized or catheter, Pop=Population, RND=Randomized, Sbj=Subject
Groups:
- BARD® LUBRI-SIL® IC Foley Catheter: Route of Administration: Urinary Bladder Catheterization
  BARD® LUBRI-SIL® IC Foley Catheter : The LUBRI-SIL® I.C. antimicrobial 100% silicone Foley catheter incorporates a formulation consisting of BACTI-GUARD®* silver alloy coating and BARD® hydrogel.
- ICET™ TIC Foley Catheter: Route of Administration: Urinary Bladder Catheterization
  ICET™ TIC Foley Catheter : The device to be evaluated in this investigation is a silver-based antimicrobial coated Foley catheter connected to an antimicrobial anti-reflux accessory (ICET Inc, Norwood, MA). The closed system is referred to as the TIC system and is designed with the objective of reducing the incidence of CAUTI. The accessory is non-tissue contacting.
Period: Overall Study
Arm/Group | BARD® LUBRI-SIL® IC Foley Catheter | ICET™ TIC Foley Catheter
Started | 46 (All randomized subjects in the Lubri-Sil arm.) | 49 (All randomized subjects in the TIC arm.)
Intent to Treat (ITT) Population | 45 (Any subject receiving the Lubri-Sil treatment after randomization.) | 46 (Any subject receiving the TIC treatment after randomization.)
Evaluable Population | 16 (Subjects w/ positive urine culture results also removed from the Lubri-Sil arm of this population.) | 14 (Subjects w/ positive urine culture results also removed from the TIC arm of this population.)
Completed | 28 | 35
Not Completed | 18 | 14
Not completed — No Treatment Received | 1 | 3
Not completed — Failed Inclusion/Exclusion | 3 | 0
Not completed — No Baseline Dips Stick & Urine Culture | 3 | 6
Not completed — No Daily Urine Sample Collected | 0 | 1
Not completed — No post-catheter sample collected | 11 | 4

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants (95 participants) includes 4 individuals who were randomized, but not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | BARD® LUBRI-SIL® IC Foley Catheter | ICET™ TIC Foley Catheter | Total
Number analyzed (Participants) | 46 | 49 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 49 | 95
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13.4) | 52.3 (16.6) | 55.6 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Prior to Study Termination; of 95 subjects randomized, 91 subjects were treated and therefore considered as part of Baseline Gender demographics.
  Participants
    Female | 24 | 30 | 54
    Male | 22 | 19 | 41
Region of Enrollment [Number; unit: participants]
  United States | 46 | 49 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Affected, During Treatment and Follow-up Time Periods, by a Catheter Associated Urinary Tract Infection (CAUTI) Event After First CAUTI Event.
Description: All randomized subjects will be followed until (1) up to 30th day from the time of catheterization or (2) the subject withdraws or is discharged from the hospital, whichever comes first and (3) 48 hours after the catheter is removed.
  Evaluable population (EP) refers to all randomized subjects successfully CZD & stayed on the CZD for ≥ 48 ± 24 hours or more without any systemic (postoperative) antibiotic for CZD/non-CZD related reasons. Subjects receiving an intercurrent course of systemic antibiotics lasting >24 hours other than surgical prophylaxis were considered non-evaluable in all analyses of effectiveness endpoints using the EP.
Time Frame: up to 30th day from the time of catheterization
Measure: Number; unit: participants
Arm/Group | BARD® LUBRI-SIL® IC Foley Catheter | ICET™ TIC Foley Catheter
Number analyzed (Participants) | 46 | 49
participants
  Number of Subject with Event | 8 | 3
  Number of Subject without Event | 37 | 43
  Number of Subjects Not Receiving Treatment | 1 | 3

2. Secondary Outcome: The Proportion of Subjects With Symptomatic Urinary Tract Infection (SUTI)
Description: Patients with catheter related SUTI are those having an indwelling urinary catheter in place at the time of specimen collection, or had an indwelling catheter within the previous 48 hours, and at least 1 of the following signs or symptoms with no other recognized cause: fever (>38°C), suprapubic tenderness, or costovertebral angle pain or tenderness and a positive urinalysis demonstrated by at least one of the following findings: a. positive dipstick for leukocyte esterase and/or nitrite, b. pyuria (urine specimen collected from the catheter with ≥10 white blood cells [WBC]/mm3 or ≥3 WBC/high power field of unspun urine), c. microorganisms seen on Gram stain of unspun urine and a positive urine
Time Frame: up to 30th day from the time of catheterization
Measure: Number; unit: Participants
Arm/Group | BARD® LUBRI-SIL® IC Foley Catheter | ICET™ TIC Foley Catheter
Number analyzed (Participants) | 46 | 49
Participants
  Number of Subjects with SUTI | 0 | 1
  Number of Subjects without SUTI | 45 | 45
  Missing - Not Assessed | 1 | 3

3. Secondary Outcome: The Proportion of Subjects With Asymptomatic Bacteremic Urinary Tract Infection (ABUTI)
Description: Patients having an indwelling urinary catheter who have no signs or symptoms (i.e., no fever (>38°C), no urgency, frequency, dysuria, suprapubic tenderness, or costovertebral angle pain or tenderness), and a positive urine culture from urine collected from the catheter sampling port (or a midstream voided clean catch urine in subjects being followed for 48 hours post catheter removal) of >105 CFU/ml with no more than 2 species of uropathogen microorganisms and a positive blood culture with at least 1 matching uropathogen microorganism to the urine culture.
Time Frame: up to 30th day from the time of catheterization
Measure: Number; unit: participants
Arm/Group | BARD® LUBRI-SIL® IC Foley Catheter | ICET™ TIC Foley Catheter
Number analyzed (Participants) | 46 | 49
participants
  Number of Subjects with ABUTI | 0 | 0
  Number of Subjects without ABUTI | 38 | 37
  Missing - Not Assessed | 8 | 12

4. Primary Outcome: The Proportion of Subjects With at Least One CAUTI
Description: CAUTI is as determined by blinded investigator assessment per protocol definition.
  DAYS TO CAUTI = (DATE OF EVENT - DATE OF CZD INSERTION) + 1. Date of event for subjects who had CAUTI is the date of urine sample collection where the CAUTI criteria are met.
  Date of event for subjects who did not have CAUTI is the last available urine culture collection date from samples collected during & post CZD.
  p-values of time of CAUTI were obtained from log-rank test. p-values of Incidence of CAUTI were obtained from the Logistic Regression Model.
  Evaluable population (EP) refers to all randomized subjects successfully CZD & stayed on the CZD for ≥ 48 ± 24 hours or more without any systemic (postoperative) antibiotic for CZD/non-CZD related reasons. Subjects receiving an intercurrent course of systemic antibiotics lasting >24 hours other than surgical prophylaxis were considered non-evaluable in all analyses of effectiveness endpoints using the EP.
  CZD = Catheterized or catheter
Time Frame: 48 ± 24 hours or more
Measure: Number; unit: participants
Arm/Group | BARD® LUBRI-SIL® IC Foley Catheter | ICET™ TIC Foley Catheter
Number analyzed (Participants) | 16 | 14
participants
  Number of Subjects With Event | 7 | 2
  Number of Subjects Without Events | 9 | 12

5. Other Pre Specified Outcome: Organism Relation to CAUTI and TIC
Description: Organisms found in relation to CAUTI events in TIC versus control.
Time Frame: up to 30th day from the time of catheterization
Measure: Number; unit: participants
Arm/Group | BARD® LUBRI-SIL® IC Foley Catheter | ICET™ TIC Foley Catheter
Number analyzed (Participants) | 46 | 49
participants
  Candida Responsible for CAUTI Events | 0 | 1
  E.Coli Responsible for CAUTI Events | 4 | 0
  Pseudomonas Responsible for CAUTI Events | 1 | 0
  Enterobacter Responsible for CAUTI Events | 1 | 0
  Klebsiella Responsible for CAUTI Events | 1 | 0
  Enterococcus Responsible for CAUTI Events | 2 | 2
  CoNS Responsible for CAUTI Events | 1 | 0
  Total Organisms Responsible for CAUTI Events | 10 | 3

ADVERSE EVENTS:
Arm/Group | BARD® LUBRI-SIL® IC Foley Catheter | ICET™ TIC Foley Catheter
Serious Adverse Events (participants affected / at risk) | 3/45 | 0/46
Other Adverse Events (participants affected / at risk) | 39/45 | 40/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BARD® LUBRI-SIL® IC Foley Catheter (N=45) | ICET™ TIC Foley Catheter (N=46)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial iscaemia (Cardiac disorders) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BARD® LUBRI-SIL® IC Foley Catheter (N=45) | ICET™ TIC Foley Catheter (N=46)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 11 (11)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 2 (2)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Gaze palsy (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (9) | 6 (6)
Tongue haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (4)
Face oedema (General disorders) | 1 (1) | 2 (2)
Infusion site extrvasation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 9 (9)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site oedema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 3 (3) | 3 (3)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 2 (2) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 2 (2)
Urine output decreased (Investigations) | 1 (1) | 1 (1)
Urine output increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 2 (2)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Brudzinski's sign (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Clonus (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 2 (2)
Monoplegia (Nervous system disorders) | 1 (1) | 1 (1)
Nystagmus (Nervous system disorders) | 3 (3) | 2 (2)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Pneumocephalus (Nervous system disorders) | 2 (2) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 4 (4)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2) | 4 (4)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Syncope (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study could not be completed for business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No